CLINICAL TRIAL: NCT01963819
Title: Therapeutic Endometrial Biopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Miacol-2013-1H
Record Dates: First submitted 2013-10-11; First posted 2013-10-16 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Infertility; Endometrium; ART; Endometrial Biopsy
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Standard treatment
- Intervention (Experimental): Endometrial biopsy before standard treatment
  Interventions: Other: Endometrial biopsy

INTERVENTIONS:
Other: Endometrial biopsy — The endometrial biopsy will be done in the luteal phase (cycle day 18-22) prior to the treatment cycle (antagonist)
  Other Names: Endometrial scratching; Endometrial injury; Local injury to the endometrium
  Arms: Intervention

SUMMARY:
The aim of this study is to evaluate the potential benefits in implantation, clinical pregnancy and live birth rates by an endometrial biopsy prior to an IVF/ICSI treatment. Including a follow up on possible pregnancy complications and data on children at birth.

Further it is planned to aspirate secretions from the uterus and take blood samples during the treatment, which presumably can provide information about the mechanisms underlying the possible effect of the treatment.

DETAILED DESCRIPTION:
Randomized controlled prospective clinical study.

ELIGIBILITY:
Inclusion Criteria:

* One or more previous failed implantation despite transfer of good quality embryons/blastocyst in a fresh IVF/ICSI treatment
* Planned Antagonist treatment
* Planned Standardized hormone treatment
* FSH: 2-12 IU/L
* Age: 18-40 years
* BMI: 18-32
* Regular menstrual cycles
* Written consent

Exclusion Criteria:

* Patients in need for a interpreter
* Suspected intrauterine abnormalities ( fibromes, polyps, adenomyosis, sactosalpinges)
* Planned use og Assisted hatching or use of specialized media
* Previous inclusion in the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Rate of clinical pregnancy | Individual outcome will be evaluated within 8 weekes after embryo transfer. Overall outcome will be evaluated after 3 years.

SECONDARY OUTCOMES:
Rate of biochemical pregnancy | Individual outcome will be evaluated within 8 weeks after embryo transfer. Overall outcome will be evaluated after 3 years.
Rate of implantation | Individual outcome will be evaluated within 8 weekes after embryo transfer. Overall outcome will be evaluated after 3 years.
Rate of live birth | Individual outcome will be evaluated within 9 months after embryo transfer. Overall outcome will be evaluated after 3 years.

OTHER OUTCOMES:
Rate of pregnancy complications | Individual outcome will be evaluated within 9 months after embryo transfer. Overall outcome will be evaluated after 3 years.
  Placenta abnormalities, pregnancy related hypetensive disorders, IUGR, GDM
Data on children and placenta at birth | Individual outcome will be evaluated within 9 months after embryo transfer. Overall outcome will be evaluated after 3 years.
  Gestationel age, Preterm birth, LGA/SGA/NGA, Gender, Placenta abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Axel Forman, MD, DMsc, Study Director — Departement of Gynaecology and Obstetrics, Aarhus University Hospital, Skejby; Inge E Agerholm, M.Sc, PhD, Principal Investigator — Fertility Clinic, Horsens Hospital; Benedicte Hauge, MD, Principal Investigator — Fertility Clinic, Horsens Hospital; Peter Humaidan, MD, DMSc, Principal Investigator — Fertility Clinic, Skive Hospital; Mia Steengaard Olesen, MD, Principal Investigator — Fertility Clinic Horsens Hospital, Aarhus University
Locations (3):
- Denmark (3):
  - Fertility Clinic, Dronninglund Hospital (Aalborg University Hospital), Dronninglund
  - Fertility Clinic, Horsens Hospital, Horsens
  - Fertility Clinic, Skive Hospital, Skive

REFERENCES:
- [Derived] Olesen MS, Hauge B, Ohrt L, Olesen TN, Roskaer J, Baek V, Elbaek HO, Nohr B, Nyegaard M, Overgaard MT, Humaidan P, Forman A, Agerholm I. Therapeutic endometrial scratching and implantation after in vitro fertilization: a multicenter randomized controlled trial. Fertil Steril. 2019 Dec;112(6):1015-1021. doi: 10.1016/j.fertnstert.2019.08.010. PMID 31843072